CLINICAL TRIAL: NCT02484963
Title: The Study of Spectrum of Sleep Disorders in Cirrhotic Patients and the Efficacy of Zolpidem in Cirrhotic Patients With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Insomnia-001
Record Dates: First submitted 2015-05-22; First posted 2015-06-30 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2016-06

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- zolpidem (Experimental): Tablet zolpidem 5mg once daily will be given for 4 weeks
  Interventions: Drug: Zolpidem
- Placebo (Placebo Comparator): One tablet of placebo will be given for 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Zolpidem
  Arms: zolpidem
Drug: placebo
  Arms: Placebo

SUMMARY:
All Cirrhosis liver patients (Child A/B/C) presenting to Institute of Liver and Biliary Sciences will be screened for sleep disturbance and excessive daytime sleepiness with Epworth sleep score/ Pittsburgh sleep quality index. 52 patients of clinical/ radiological/ biopsy proven cirrhosis (Child A/B) will be enrolled after ruling out possibility of psychiatric illnesses like depression and anxiety with the help of PHQ-9 / GAD-7 questionnares. Patients who are suffering with sleep disturbance as evaluated with Pittsburgh sleep quality index will undergo polysomnography and will be randomised to two groups after fulfilling all inclusion criterias. Patients in group (Group 1) will receive zolpidem 5mg at bed time daily and patients in control group will receive placebo at bed time daily. The treatment will be continued for 4 weeks. After 4 weeks enrolled patients will be reassessed with PSQI and polysomnography. All patients will be advised regarding sleep hygiene.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Clinical, Biochemical, Radiological ,Histological evidence of cirrhosis of all etiology
* Child A and B cirrhosis (for intervention part)
* Cirrhosis patients giving h/o persistent sleep disturbances (PSQI≥5)
* Child A, B and C cirrhosis (for observational part)

Exclusion Criteria:

* Active alcohol intake or intake within 1 month of enrollment
* Active substance abuse or intake within 1 month of enrollment
* Known psychiatric and neurological disorders
* Patient using antidepressant, anticonvulsants, other hypnotics
* Pregnancy or lactation
* Overt hepatic encephalopathy (grade 2,3,4)
* Child C cirrhosis (for intervention part)
* Acute decompensated state of CLD (Chronic Liver Disease) - GastroIntestinal bleed, increased jaundice, HE (Hepatic Encepahlopahty) , SBP (Spontaneous Bacterial Peritonitis).
* HCC (HepatoCellular Carcinoma) with portal vein thrombosis
* Acute febrile illness/ acute infection
* Post TIPS (Transjugular Intrahepatic Portosystemic shunt)patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Improvement in quality of sleep in CHILD A/B cirrhosis patients after 4 weeks as measured by total sleep time | 4 weeks

SECONDARY OUTCOMES:
Precipitation of Hepatic encephalopathy with Zolpidem | 4 weeks
Increase in daytime sleepiness with zolpidem as measured by ESS | 4 weeks
Improvement in sleep efficiency after treatment | 4 weeks
Reduction in periodic limb movements after treatment | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India